CLINICAL TRIAL: NCT05256836
Title: Effects of Tablet Computer-based Cognitive Training in Patients With Idiopathic REM Sleep Behavior Disorder
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment suspended
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2105-117-1220
Record Dates: First submitted 2022-02-06; First posted 2022-02-25 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tablet group (Experimental): A total of 36 sessions per week for 12 weeks of cognitive training program using a tablet computer are performed.
  Interventions: Other: Tablet computer-based cognitive training program
- control group (No Intervention): Subjects assigned to the control group did not receive any separate cognitive training for 12 weeks.

INTERVENTIONS:
Other: Tablet computer-based cognitive training program — The subject of the study executes a program mounted on a tablet personal computer (PC) (Samsung Galaxy Tab S6 Lite) and performs a cognitive training task by touching the screen with the index finger.
  It consists of 10 tasks related to the activity of daily living: 1) taking medicine, 2) making a phone call, 3) taking a shower, 4) doing laundry, 5) finding directions, 6) riding the bus, 7) buying goods, 8) Money management, 9) ingredient sorting, 10) meal preparation.
  It is involved in cognitive functions in various domains such as attention, working memory, processing speed, problem solving, visuospatial ability, verbal and visuospatial memory.
  There are three levels of difficulty for each task, high, medium, and low, and the difficulty becomes more difficult as session 1 to 36 progresses.
  One cognitive training session lasts about 30 minutes.
  Arms: tablet group

SUMMARY:
To evaluate the effectiveness of tablet computer-based cognitive training in patients with idiopathic REM sleep behavior disorder.

DETAILED DESCRIPTION:
Rapid eye movement (REM) sleep behavior disorder (RBD) is a parasomnia characterized by abnormal movement to reproduce dreams and loss of skeletal muscle tension during REM sleep. Idiopathic RBD (iRBD) refers to the absence of any predisposing factors or comorbid neurological disorders. iRBD is considered the prodromal stage of alpha-synucleinopathy.

Through past studies, it has been confirmed that cognitive function decline has already occurred in a significant number of iRBD patients. However, there is still no treatment that can suppress or delay the onset of neurodegenerative diseases.

The cognitive function improvement effect of computerized cognitive training in the elderly and patients with mild cognitive impairment is known. However, the effect of cognitive training on improving cognitive function in iRBD patients has not been studied.

The investigators developed a program that allows patients to train cognitive functions in various domains by repeatedly performing tasks related to daily life activities. In addition, by loading the program on the tablet computer, it is possible to participate in the training easily at home using the touch screen without visiting the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60-80 years old who have been diagnosed with iRBD through nocturnal polysomnography according to the International Classification of Sleep Disorders 3rd Edition (ICSD-3) diagnostic criteria
* Those who gave their written consent to participate in the study

Exclusion Criteria:

* Patients with neurodegenerative diseases including Parkinson's disease, dementia, and multiple system atrophy
* Patients with secondary causes of RBD
* Patients with severe hearing, visual impairment, or motor impairment
* Patients who have received cognitive training within the last year

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Korean version of the Consortium to Establish a Registry for Alzheimer's Disease Assessment Packet (CERAD-K) total score | Change from baseline CERAD-K total score at 12 weeks
  Z score of total 5 domains (attentive, memory, language, visuospatial and executive functions)

SECONDARY OUTCOMES:
Change in CERAD-K attention score | Change from baseline CERAD-K attention score at 12 weeks
  Scores for each of the 5 domains
  1.Attention
  * Trail making test A (0~360): higher scores mean a worse outcome
  * Stroop test (word) (0~): higher scores mean a better outcome
Change in CERAD-K memory score | Change from baseline CERAD-K memory score at 12 weeks
  Scores for each of the 5 domains 2.Memory
  * Word registration (0~30): higher scores mean a better outcome
  * Word recall (0~10): higher scores mean a better outcome
  * Word recognition (0~10): higher scores mean a better outcome
  * Constructional recall (0~11): higher scores mean a better outcome
Change in CERAD-K language score | Change from baseline CERAD-K language score at 12 weeks
  Scores for each of the 5 domains 3.Language
  - Boston naming test (0~15): higher scores mean a better outcome
Change in CERAD-K visuospatial function score | Change from baseline CERAD-K visualspatial function score at 12 weeks
  Scores for each of the 5 domains 4.Visuospatial function
  - Constructional behavior (0~11): higher scores mean a better outcome
Change in CERAD-K executive function score | Change from baseline CERAD-K executive function score at 12 weeks
  Scores for each of the 5 domains 5.Executive function
  * Trail making test B (0~300): higher scores mean a worse outcome
  * Language fluency (0~): higher scores mean a better outcome
  * Stroop test (word/color) (0~): higher scores mean a better outcome
Change in mini-mental status examination in the Korean version (MMSE-K) score | Change from baseline MMSE-K score at 12 weeks
  minimum value: 0, maximum value: 30 (higher scores mean a better outcome)
Change in Korean version of Montreal Cognitive Assessment (MoCA-K) score | Change from baseline MoCA-K score at 12 weeks
  minimum value: 0, maximum value: 30 (higher scores mean a better outcome)
Change in resting electroencephalography (EEG) power spectrum | Change from baseline EEG power spectrum at 12 weeks
  distribution of power into frequency components composing the signal (delta, theta, alpha, beta)
Change in resting electroencephalography (EEG) weighted phase lag index | Change from baseline EEG weighted phase lag index at 12 weeks
  a functional connectivity measure that quantified how consistently 90° (or 270°) phase 'lagging' one EEG signal was compared to another (From 0 to 1, if it is close to 1, the connectivity is high)
Change in event-related potential (ERP) reaction time | Change from baseline ERP reaction time at 12 weeks
  time (ms) from target presentation to button press
Change in event-related potential (ERP) hit rate | Change from baseline ERP hit rate at 12 weeks
  the probability that an old item is either correctly recognized, or not
Change in event-related potential (ERP) N2 amplitude | Change from baseline ERP N2 amplitude at 12 weeks
  The N2 peak (μV) is a fronto-central maximal negativity observed approximately 150-400 ms after stimulus onset
Change in event-related potential (ERP) time-frequency analysis | Change from baseline ERP time-frequency analysis at 12 weeks
  Indicates the power of the EEG frequency at a specific time

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Young Jung, professor, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea